CLINICAL TRIAL: NCT03172650
Title: Effect of Non-alcoholic Fatty Liver Disease on Kidney Functions: Observational Case Control Study in Upper Egypt
Brief Title: Effect of Non-alcoholic Fatty Liver Disease on Kidney Functions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: NAFLD
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Glomerular Filtration Rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: non alcoholic fatty liver disease patients
  Interventions: Diagnostic Test: glomerular filtration rate
- Control group: fatty liver patients
  Interventions: Diagnostic Test: glomerular filtration rate

INTERVENTIONS:
Diagnostic Test: glomerular filtration rate — collection of blood sample 5 milliliter for calculation of glomerular filtration rate

SUMMARY:
Non-alcoholic fatty liver disease is the most common cause of chronic liver disease worldwide. It is defined as the accumulation of fat (>5%) in the liver cells in the absence of excessive alcohol intake or other causes of liver disease including viral, drug-induced, or autoimmune. Non-alcoholic fatty liver disease is a hepatic manifestation of metabolic syndrome.

ELIGIBILITY:
Inclusion criteria:

* All non alcoholic fatty liver disease patients evidenced by abdominal ultrasound.
* Urine analysis whether normal or renal sedimentation.

Exclusion criteria:

1. Alcoholic fatty liver patients.
2. patients known to have diabetes mellitus.
3. patients with other causes of liver disease as viral hepatitis, drug induced,or autoimmune.
4. patients known to have kidney disease.
5. Hypertension.
6. Hyperuricemia.
7. Impaired urea and creatinine patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited outpatient clinic of internal medicine of Luxor international hospital and Assiut university hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with abnormal laboratory glomerular filtration rate | 1 day
  decreased glomerular filtration rate <60 mL/minute will be considered abnormal

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No